CLINICAL TRIAL: NCT07373743
Title: Pharmacokinetic (PK) Study of Tafenoquine in Healthy Adults
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2026-01-UMU; PR241374 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2026-01-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetic in Normal Population
Keywords: Tafenoquine; CYP2D6; Pharmacokinetic
MeSH Terms: interventions — tafenoquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Normal Metabolizers (NM) (Experimental): Participants with normal CYP2D6 enzyme activity receiving a single 450 milligram (mg) dose of tafenoquine.
  Interventions: Drug: Tafenoquine Oral Tablet
- Intermediate Metabolizers (IM) (Experimental): Participants with decreased activity of the enzyme leading to variable effects i.e., either no effect, increased adverse effects from TQ or reduced efficacy of the drug in endemic areas due to inadequate metabolism receiving a single 450mg dose of tafenoquine.
  Interventions: Drug: Tafenoquine Oral Tablet
- Poor Metabolizers (PM) (Experimental): Participants with no enzyme activity at all, leading to a null phenotype and no drug metabolism receiving a single 450mg dose of tafenoquine.
  Interventions: Drug: Tafenoquine Oral Tablet

INTERVENTIONS:
Drug: Tafenoquine Oral Tablet — Single, 450mg dose

SUMMARY:
The goal of this clinical trial is to learn how people's different genetic makeups affects how their bodies convert the FDA approved drug ARAKODA (tafenoquine) to its active form. Tafenoquine is a drug that is taken to prevent malaria for people traveling to areas where there is malaria. This trial will be in healthy participants age 18-65.

DETAILED DESCRIPTION:
This trial will explore the how different CYP450 2D6 phenotypes metabolize a single 450mg dose of tafenoquine. Pharmacokinetic (PK) blood and urine samples, and research samples will be obtained at specific timepoints during the 2-month study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 at the time of consent, weighing between 132 and 250 pounds
2. Ability and willingness to sign informed consent
3. Available for the study period
4. Willing to use contraception for the duration of the study
5. Agree not to take over the counter antioxidants, vitamin C or vitamin E, 2 weeks prior to dosing and 7 days post dosing

Exclusion Criteria:

1. Women: positive urine pregnancy test at screening or day of dosing
2. Women who are lactating or intend to become pregnant during the study period.
3. Acute or chronic clinically significant hematologic, pulmonary, cardiovascular, hepatic, or renal functional abnormality as determined by medical history, physical examination or laboratory screening.
4. History of allergic reaction to tafenoquine or primaquine.
5. Scheduled receipt of any vaccine 1 week prior to or after 4 weeks tafenoquine dosing. Routine COVID and influenza vaccination will be allowed outside of this timeframe.
6. Currently taking metformin, dofeltilide or other medication with known multidrug and toxin extrusion enzyme (MATE) metabolism.
7. Known or suspected congenital or acquired immunodeficiency; or receipt of immunomodulation therapy such as anti-cancer chemotherapy or radiation therapy.
8. Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the participant from participating in the study.
9. Participants with hemoglobin, Creatinine, BUN, Albumin, eGFR; ALT, and AST of grade 2 or greater. Any exclusionary lab abnormality may be repeated once. If a repeat screening blood test is performed, only the result of the second test will be reviewed and used to determine eligibility.
10. G6PD result not normal or < 70% activity
11. Significant screening physical examination abnormalities or chronic medical condition that in the opinion of the investigator may impact participant safety, including BMI > 35kg/m2
12. Participation (active or follow-up phase) or planned participation in another vaccine, or drug, in the 4 weeks prior to or during the trial
13. Beliefs that bar the administration of blood products or transfusions
14. Clinician discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Tafenoquine levels in blood over time | Pre-dose, 4, 8, 12, and 24 hours (Day 2) and Days, 3, 4, 5, 6, 7, 8, 15, 22, 29, and 57.
Tafenoquine levels in urine over time | Pre-dose, total volume collected between 0-4, 4-8, 8-12, 12-24 hours and then single void collections on Days 3, 4, 5, 6, 7, 8, 15, 22, 29, 57.

SECONDARY OUTCOMES:
Methemoglobin Levels | Pre-dose, 4, 8, 12, and 24 hours (Day 2) and Days, 3, 4, 5, 6, 7, 8, 15, 22, 29, and 57
  Methemoglobin Levels at defined PK timepoints
Laboratory abnormalities | Pre-dose, Day 4 and 15
  Complete Blood Count and reticulocyte count
Adverse Events | From Day 1 to Day 29
Serious Adverse Events | Day 1 to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spring, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Upstate Global Health Institute, East Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies the primary results in a publication.
Time Frame: IPD will be shared with the primary publication
Access Criteria: Primary IPD will be published with the primary manuscript describing the study. Requests for additional information can be requested by emailing warel@upstate.edu.